CLINICAL TRIAL: NCT03948074
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Crossover N-of-1 Study Design of the Use of Medicinal Cannabis Oil-Based Extracts for Symptom Management in Cancer Patients
Brief Title: Cannabis For Cancer-Related Symptoms
Acronym: CAFCARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pippa Hawley (Other)
Responsible Party: Sponsor-Investigator, Pippa Hawley, Division Head of Palliative Care, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFCARS
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pain; Nausea; Anxiety; Sleep Disturbance
MeSH Terms: conditions — Pain; Nausea; Anxiety Disorders; Parasomnias | interventions — nabiximols; Dronabinol; Cannabidiol

STUDY DESIGN:
Intervention Model Description: An N-of-1 trial is a crossover trial, usually randomized and often blinded, conducted in a single patient. This type of trial provides an objective, data-driven way to determine the most effective intervention for an individual patient from among a set of competing interventions and to investigate the side-effect profiles of each intervention.
  It is possible to analyze the results produced by each N-of-1 trial in a series separately in order to determine whether (i) the active treatment(s) involved in the trial were effective for the corresponding patient or (ii) the novel treatment(s) involved in the trial were effective relative to the established treatment. It is also possible to aggregate the results produced by a series of simultaneous N-of-1 trials (all conducted in a similar way) using either meta-analytic methods or mixed effects modelling in order to obtain information on how to treat subsets of the target patient population or even the entire patient population at large.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High THC/Low CBD Cannabis Oil (Experimental): THC+THCa = 573 mg CBD+CBDA = 0 mg Total cannabinoids = 573 mg (0.95mg/drop) Dried marijuana equivalent = 5g
  Interventions: Drug: Cannabis
- Low THC/High CBD Cannabis Oil (Experimental): THC+THCa = 37mg CBD+CBDA = 784mg Total cannabinoids = 821mg (1.37mg/drop) Dried marijuana equivalent = 6g
  Interventions: Drug: Cannabis
- Equal amounts of THC/CBD Cannabis Oil (Experimental): THC+THCa = 516mg CBD+CBDA = 456mg Total cannabinoids = 972mg (1.62mg/drop) Dried marijuana equivalent = 6g
  Interventions: Drug: Cannabis
- Placebo Oil (Placebo Comparator): Medium Chain Triglyceride (MCT) oil
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Medicinal Cannabis Oil
  Other Names: Tetrahydrocannabinol; Cannabidiol

SUMMARY:
Clinical evidence is urgently needed to be able to advise patients on which cannabis-based products to take, or to avoid, in managing cancer-related symptoms. This trial was therefore designed to determine which cannabis extract combination (High THC-Low CBD, Low THC-High CBD, or Equal amounts of THC and CBD) is most effective at treating cancer related symptoms for each patient relative to placebo. Investigators propose a randomized, double-blind, N-of-1 trial to test the effectiveness of each cannabis extract combination using cannabis oils in a minimum of 120 patients on 4 cancer-related symptoms: nausea, pain, anxiety and sleep disturbance.

The three active treatments will be the following cannabis oil extract combinations: High THC/Low CBD, Low THC/High CBD, and Equal amounts of THC/CBD.

* THC = Tetrahydrocannabinol
* CBD = Cannabidiol

The placebo treatment will be Medium Chain Triglyceride (MCT) oil. The active oils and the placebo are similar in taste, smell and effectively blind subjects.

Primary objective:

To identify whether there is an active cannabis extract that is more effective than placebo in managing overall cancer-related symptoms for individual subjects who completed at least 1 treatment cycle for the entire patient population represented by those individual subjects, and for subsets of that subject population defined by relevant baseline patient characteristics.

Secondary objective:

To identify whether there is a cannabis extract that is more effective than placebo in managing each of the 4 index symptoms (pain, nausea, anxiety and sleep disturbance) for individual subjects who completed at least 1 treatment cycle, for the entire patient population represented by those individual subjects, and for subsets of that subject population defined by relevant baseline patient characteristics.

Tertiary objectives:

To investigate the safety (e.g., serious adverse events) of each of the three cannabis extracts.

To identify subject preference of each of the 4 oils (if any).

DETAILED DESCRIPTION:
Investigators propose a study consisting of a series of N-of-1 trials comparing 3 different active cancer-related symptom management treatments against a placebo treatment in terms of effectiveness and safety. Using formal statistical modeling, effectiveness will be assessed for single patients, for the entire patient population and for relevant subsets of the patient population defined by baseline patient characteristics. Safety will be assessed in a descriptive fashion for all patients who are part of the safety population.

Subjects will be on treatment in the study for a minimum of 16 days with the opportunity to repeat the 16-day cycle of cancer-related symptom treatment with all four oil extracts up to 2 more times. The extracts will be supplied to subjects at the beginning of the study in four distinct 30-ml bottles, randomly labelled as #1, #2, # 3 and # 4. The random labelling will be generated via a computer-generated randomization code.

The study will include at least 120 adult subjects (recruitment target 150 to allow for drop-outs) residing in Canada who have symptoms from cancer and/or from cancer treatment but will exclude patients with active recreational use, cannabis use disorder, or high risk of diversion.

Each treatment cycle will have a length of 16 days and will consist of 4 four-day periods. The first 2 days of each 4-day period will be a washout period where data will not be used for the analysis of effectiveness, to make sure there is no confusion with effects from the prior period. Subjects can use one and only one cannabis oil extract during each period to treat their cancer-related symptom(s).

Given a cannabis oil extract, the daily use of that extract by patients will involve the following: On each day within a specific treatment cycle, the patient will be asked to take a minimum of 3 drops of that extract per day (e.g., in the morning) and if any of the four major symptoms (nausea, pain, anxiety, and sleep disturbance) continue to trouble the patient as the day progresses, they will be instructed to take up to 3 drops every 4 hours for a maximum of 6 times a day (for a total of no more than 18 drops per day).

All subjects will be instructed to use the following validated scales: Edmonton Symptom Assessment Scale (ESAS) and Patients' Global Impression of Change Scale (PGIC). The revised ESAS will be used modified to include sleep disturbance (previously validated), and added night sweats in replacement of the additional symptom option (ESAS-r-SN) because of reports of benefit of medical cannabis for this symptom and its relevance for sleep disturbance.This is in order to capture a complete picture of potential factors contributing to sleep disturbance. Additionally, subjects will be instructed to fill in a study medication use log which will record the timing and dose of each extract applications, any side effects associated with each application, as well as any rescue medication (if taken).

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years of age;
* Competent to consent to participation in the study;
* Must have at least one of the following cancer-related symptoms or a cancer treatment-related symptoms which is causing distress: Nausea; Pain; Anxiety; Sleep Disturbance; (based on ESAS-r-SN score ≥4/10)
* Symptom(s) are expected to be stable throughout the duration of the study;
* Expecting to live for at least 4 months;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2;
* Willing to commit to not taking cannabis in any form other than the study products for the duration of the study;
* Able to reliably communicate with the research team, either directly or through a translator;
* Accessible by telephone.

Exclusion Criteria:

* Their current symptoms are not related to cancer or cancer treatment;
* They have a current cannabis or other substance dependence or misuse disorder as defined by the revised Cannabis Use Disorder Identification Test (CUDIT-R) score of 8 or above;
* They admit to cannabis use for any purpose (recreational or medicinal) more than once a week during the month prior to study entry;
* They have a history of psychosis with, or other intolerance to cannabis or cannabinoids;
* They have an active psychiatric disorder likely, in the investigator's opinion, to interfere with adherence to study protocol;
* They have any concurrent condition likely to interfere with completion of the study protocol, such as allergy to any component of the study products;
* They are pregnant or planning to get pregnant or they are lactating females;
* They are women of childbearing potential (<2 years after last menstruation) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal);
* They have reproductive potential and fail to use adequate birth control;
* They are on another clinical trial or expect to start one prior to study completion;
* They have oral disease which might impair trans-mucosal absorption, e.g. oral mucositis;
* They are taking medications that might be affected by an interaction with cannabinoids in a clinically significant manner (CYP1A1, 1A2, and 1B1) and cannot be switched to a different medication;
* They live in an environment with high risk of theft or diversion of study products;
* They have a concurrent condition that requires changes to current medications within the 48 days on study treatment.
* They have serious cardiovascular disease such as ischemic heart disease, including arrhythmias, poorly controlled hypertension, severe heart failure, recent (within 6 months) MI.
* They have first degree relatives with schizophrenia.
* They have history of epilepsy or repeated seizures or brain metastases.
* They are unable or unwilling to refrain from operating heavy machinery for the duration of their participation in this study.
* They are unable or unwilling to refrain from consuming alcohol for the duration of their participation in this study.
* They expect to leave Canada during the study period, as the study products cannot be taken across any international border (land, sea or air).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Average Patients' Global Impression of Change (PGIC) for overall cancer-related symptoms | 16-48 days; 90 minutes after each dose
  The PGIC provides a single, general estimate of improvement or deterioration using scores from 1 to 7 and has been used as a research outcome indicator in a variety of contexts, particularly in chronic pain.
  The PGIC asks subjects to rate their current status as:
  1. No change (or condition worse)
  2. Almost the same (hardly any change at all)
  3. A little better (no noticeable change)
  4. Somewhat better (change has not made any real difference
  5. Moderately better (slight but noticeable change)
  6. Better (definite improvement that has made a real and worthwhile difference)
  7. A great deal better and a considerable improvement that has made all the difference
  Subjects will be reporting their PGIC score 90 minutes after each dose of cannabis oil (1 to 6 times daily). Only scores collected on non-washout days of a treatment cycle corresponding to a particular oil formulation will be used.

SECONDARY OUTCOMES:
Average change from baseline in the Edmonton Symptom Assessment System - revised to include Sleep Disturbance and Night Sweats (ESAS-r-SN) score | 16-48 days; once daily
  The ESAS-r-SN is a set of 0-10 numerical scales that patients use to rate the severity of the most common cancer-related symptoms. A score of 0 means that patients are not experiencing that symtpom and a score of 10 indicates that patients are experiencing the most severe symptom (for example, experiencing a pain score of 10 indicates worst possible pain).
  Subjects will be reporting their ESAS-r-SN scores once daily. Only scores collected on non-washout days of a treatment cycle corresponding to a particular oil formulation will be used.

OTHER OUTCOMES:
Percent of subjects who prefer each study oil (Oil 1, 2, 3 or 4) | 16-48 days
  Subjects will be asked by study personnel at the end of the study which oil they preferred most (i.e. Oil 1, 2, 3, or 4) after study completion but prior to un-blinding and preference of oils will be recorded. Percentages of subjects who prefer each type of oil will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Hawley, FRCPC, Principal Investigator — BC Cancer
Locations (8):
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Center of the North, Prince George, British Columbia
  - BC Cancer Vancouver, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Kingston Health Sciences Centre - Kingston General Hospital Site, Kingston, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Santé Cannabis, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No